CLINICAL TRIAL: NCT00341289
Title: Environmental and Behavioral Risk Factors for Childhood Drowning
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903141; 03-CH-N141
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-09-02

CONDITIONS: Drowning
Keywords: Submersion; Epidemiology; Fatal; Child; Swim; Drowning; Survey
MeSH Terms: conditions — Drowning

SUMMARY:
This study will examine the relationship between swimming lessons, swimming ability, and other risk factors or protective factors, and the risk of drowning among children. The study's primary focus is on children between 1 and 4 years of age, with a secondary focus on older children up to 19 years of age. Drowning is the second leading cause of accidental death among children under 5 years of age, with drowning rates peaking among 1- to 2- year-olds.

The study will examine the circumstances of cases of children between 1 and 19 years of age who have drowned in a body of water where swimming ability might have been a risk factor, such as a pool, Jacuzzi, hot tub, pond, lake, river, canal quarry, irrigation ditch, dam, or ocean. (Drowning is defined as death from asphyxia while submerged, or within 24 hours of the submersion.)

The victims' parents or guardians will be interviewed about their child's general health, temperament, motor development, swimming ability, history of swimming lessons, and exposure to water. In addition, they will be asked about environmental factors related to the child's drowning, such as if a lifeguard was present or if, in the case of a pool drowning, there was a fence around the pool. They will be asked about parental norms regarding child supervision and pool-provider advice regarding swimming instruction. Parents of older children will be asked about their child's risk-taking and sensation-seeking behaviors. Information on additional risk factors, such as the remoteness of the site of the drowning and the victim's blood alcohol level will also be obtained.

The above information will be compared with similar information gathered from parents of control subjects-that is, children who are the same age as the victims and who live in the same geographic area. For adolescent cases, information about swimming in unguarded sites or drinking alcoholic beverages while in or around water will be obtained from direct interviews with adolescents, as parents may not have accurate information in these areas.

The information gained from this study will provide guidance for the development of interventions to prevent childhood drowning.

DETAILED DESCRIPTION:
Drowning is the second leading cause of unintentional injury death among children in the United States. Children under five years of age are at particularly increased risk with drowning rates peaking among 1-2 year olds. While some preventive strategies, such as pool fencing, are known to be effective, the impact of other preventive strategies is unclear. For example, data regarding the relationship between swimming lessons or swimming ability and the risk of drowning are lacking, making it difficult to formulate guidelines and policies about enrollment of young children in swimming lessons. Information about risk and protective factors for childhood drownings will provide valuable guidance for the design of future interventions to prevent these tragic deaths.

This study utilizes a case-control design to evaluate the relationship between swimming lessons, swimming ability, and other risk or protective factors on the one hand, and the risk of drowning on the other. The primary study hypothesis addresses the relationship between swimming lessons and the risk of drowning among children ages 1 to 4 years, while secondary hypotheses address risk and protective factors for drowning among older children. Parents or guardians of drowning victims and parents/guardians of age-matched controls will be interviewed. A short interview will also be conducted with adolescent controls, aged 14-19 years. Interviews include questions regarding exposure to water, swimming ability, participation in swimming lessons, and a number of other factors that might influence the risk of drowning.

Cases will be identified through a consortium of medical examiners/coroners (ME/C). As part of the investigation of drowning deaths, investigators from the medical examiners/coroners' offices routinely collect information about the circumstances surrounding the death; however, the format and content varies somewhat with jurisdiction. In the first phase of the proposed study a consortium of ME/C's will be assembled and a short abstract form will be developed to standardize collection of information relevant to the investigation. At the conclusion of the routine investigation, the investigator from ME/C office will introduce the current study to the parent/guardian. Case families, who have not indicated a refusal for a telephone interview, will be contacted by study staff for a more in-depth interview. Random digit dialing (RDD) will be used to identify appropriately matched control children. Study interviews will be conducted by telephone.

ELIGIBILITY:
* INCLUSION CRITERIA - CASES:

Drowning in which the submersion event occurred during the study period. Drowning is defined as death from asphyxia due to submersion in a liquid medium.

Age: Greater than or equal to 12 months and less than 20 years at the time of the event.

Site of submersion: Open body of water (such as a pool, Jacuzzi, hot tub, pond, lake, river, canal, quarry, irrigation ditch, dam, or ocean).

Place of residence: Cases and their parent/guardian must be residents of the United States.

EXCLUSION CRITERIA - CASES:

Ice Water Submersions, submersions that are intentional or suspected of being intentional, motor vehicle related drownings, submersions in bathtubs, toilets, sinks, or buckets.

For bodies of water that do not easily fit into the above categories, inclusion will be restricted to bodies of water where swimming ability might be related to the risk of drowning.

INCLUSION CRITERIA - CONTROLS:

Controls will be children, who have not experienced a serious submersion event (as defined above), and who reside in the same geographic area as cases.

Greater than or equal to 12 months and less than 20 years on the reference date (date of submersion for matched case).

Place of residence: Controls and their parent/guardian must reside in the United States and will be matched to cases by county of residence.

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1430
Dates: Start 2003-03-17; Primary Completion 2007-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), 9000 Rockville, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gulaid JA, Sattin RW. Drownings in the United States, 1978-1984. MMWR CDC Surveill Summ. 1988 Feb;37(1):27-33. No abstract available. PMID 3127683
- [Background] Quan L, Gore EJ, Wentz K, Allen J, Novack AH. Ten-year study of pediatric drownings and near-drownings in King County, Washington: lessons in injury prevention. Pediatrics. 1989 Jun;83(6):1035-40. PMID 2726330
- [Background] Wintemute GJ. Childhood drowning and near-drowning in the United States. Am J Dis Child. 1990 Jun;144(6):663-9. doi: 10.1001/archpedi.1990.02150300061018. PMID 2189297